CLINICAL TRIAL: NCT04712344
Title: Randomized Controlled Phase 2b Clinical Study in Parallel Groups for the Assessment of Efficacy and Safety of Therapy With COVID-19 Convalescent Plasma Plus Standard Treatment vs. Standard Treatment Alone of Subjects With Severe COVID-19
Brief Title: Assessment of Efficacy and Safety of Therapy With COVID-19 Convalescent Plasma in Subjects With Severe COVID-19 (IPCO)
Acronym: IPCO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKER-COV2-01
Record Dates: First submitted 2020-12-30; First posted 2021-01-15 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Severe COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Serotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 convalescent plasma (Experimental): A total of three units of COVID-19 convalescent plasma administered on three separate occasions during Day 1 and Day 2 and standard treatment.
  Interventions: Biological: COVID-19 convalescent plasma
- Standard treatment (No Intervention): Standard treatment.

INTERVENTIONS:
Biological: COVID-19 convalescent plasma — Infusion of a total of three units of COVID-19 convalescent plasma administered on three separate occasions during Day 1 and Day 2 in Addition to standard treatment.
  Arms: COVID-19 convalescent plasma

SUMMARY:
This phase 2b clinical study will enroll adult subjects of both sexes with ARDS due to COVID-19 necessitating invasive mechanical ventilation.

DETAILED DESCRIPTION:
The primary objective of the study is the assessment of impact of immune therapy with COVID-19 convalescent plasma on severity of COVID-19.

The secondary objectives is the Impact of immune therapy with COVID-19 convalescent plasma on markers for ARDS due to severe COVID-19 infection; short-term all-cause mortality; time course of ARDS due to severe COVID-19 and assessment of safety and tolerability of immune therapy with COVID-19 convalescent plasma.

As a primary endpoint/variable we will assess change in SOFA score from Baseline Visit to Day 8.

The study design will be prospective, open-label, randomized, controlled and parallel-grouped.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subject aged ≥18 years.
2. Estimated BMI ≥19kg/m² to ≤40kg/m².
3. Florid1 SARS-CoV-2 infection confirmed by RT-PCR in tracheo-bronchial secretion sample or pharyngeal swab sample.
4. ARDS with Horovitz index <300mmHg.
5. Necessity of invasive mechanical ventilation.
6. Written informed consent obtained from the subject's legal representative or under such arrangement as is legally acceptable in Germany (
7. Subject's assent if obtainable

Exclusion Criteria:

1. Previous exposure to COVID-19 convalescent plasma.
2. Adverse reaction to plasma proteins in medical history.
3. Interval >72h since endotracheal intubation.
4. Current or imminent necessity of ECMO treatment.
5. Pre-existing COPD GOLD stage 4.
6. Chronic congestive heart failure NYHA ≥3.
7. Pre-existing left ventricular ejection fraction <30%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in SOFA score from Baseline Visit | [Day 1, Visit 2] to Day 8 [Visit 9]
  Change in Sequential organ failure assessment (SOFA) score predicts Predicts ICU mortality based on lab results and clinical data. SOFA includes PaO2, the Glasgow Coma Scale, Mean arterial pressure OR Administration of sedatives, Bilirubin(mg/dl), Creatinine (mg/dl) and platelets. All values are rated with a value of 1 to 4 (worst condition) and are added up gradually to a final score. The lower the SOFA score, the better is the prognosis (Maximum value 24)

SECONDARY OUTCOMES:
Assessment of impact of immune therapy with COVID-19 convalescent plasma on markers for ARDS due to severe COVID-19 infection | Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15]
  Mean number of days without invasive mechanical ventilation during the period from Baseline Visit [Day 1, Visit 2] until and including Day 8 [Visit 9], Day 15 [Visit 13], and Day 29 [Visit 15], per treatment group and per subject.
  Time from Baseline Visit [Day 1, Visit 2] to extubation.
Assessment of impact of immune therapy with COVID-19 convalescent plasma on short-term all-cause mortality | Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15]
  Assessment of mortality during defined time-frame
Assessment of impact of immune therapy with COVID-19 convalescent plasma on oxygen supply in patients with ARDS due to severe COVID-19 | Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15]
  Number of subjects without supplemental oxygen on Day 8 [Visit 9], on Day 15 [Visit 13], and on Day 29 [Visit 15].
Assessment of impact of immune therapy with COVID-19 convalescent plasma on oxygen demand in patients with ARDS due to severe COVID-19 | Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15]
  Proportion of subjects without supplemental oxygen on Day 8 [Visit 9], on Day 15 [Visit 13], and on Day 29 [Visit 15].
Assessment of impact of immune therapy with COVID-19 convalescent plasma on Duration of Oxygen supply in patients with ARDS due to severe COVID-19 | Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15]
  Mean number of days without supplemental oxygen during the period from Baseline Visit [Day 1, Visit 2] until and including Day 8 [Visit 9], Day 15 [Visit 13], and Day 29 [Visit 15], per treatment group and per subject.
Assessment of impact of immune therapy with COVID-19 convalescent plasma on PEEP in patients with ARDS due to severe COVID-19 | Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15]
  Mean relative change of PEEP from Baseline Visit [Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15] or until stop of invasive mechanical ventilation, whichever comes first.
Assessment of impact of immune therapy with COVID-19 convalescent plasma on FiO2 in patients with ARDS due to severe COVID-19 | Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15]
  Mean relative change of FiO2 from Baseline Visit [Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15] or until stop of invasive mechanical ventilation, whichever comes first.
Assessment of impact of immune therapy with COVID-19 convalescent plasma on driving pressure in patients with ARDS due to severe COVID-19 | Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15]
  Mean relative change of driving pressure from Baseline Visit [Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15] or until stop of invasive mechanical ventilation, whichever comes first.
Assessment of impact of immune therapy with COVID-19 convalescent plasma on Duration of invasive mechanical Ventilation in patients with ARDS due to severe COVID-19 | Day 1, Visit 2] to all subsequent visits until and including Day 29 [Visit 15]
  Time from Baseline Visit [Day 1, Visit 2] to stop of invasive mechanical ventilation.

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Willam, MD, Principal Investigator — University Hospital Erlangen
Locations (1):
- University Hospital Erlangen, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No